CLINICAL TRIAL: NCT03774576
Title: A Non-Randomized, Open Label, One Sequence, Two-Period Cross-Over Study to Investigate the Effect of CYP3A Inhibition on the Pharmacokinetics of RO7017773 in Healthy Participants
Brief Title: A Study to Investigate the Effect of CYP3A Inhibition on the Pharmacokinetics of RO7017773 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP40822; 2018-002889-40 (EudraCT Number)
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Results first posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RO7017773 (Experimental): Single dose of RO7017773
  Interventions: Drug: RO7017773
- RO7017773 and Itraconazole (Experimental): Single dose of RO7017773 and multiple doses of itraconazole
  Interventions: Drug: RO7017773; Drug: Itraconazole

INTERVENTIONS:
Drug: RO7017773 — Single doses of RO7017773
Drug: Itraconazole — Multiple doses of Itraconazole
  Other Names: Sporanox
  Arms: RO7017773 and Itraconazole

SUMMARY:
The purpose of this study is to investigate the effect of multiple oral doses of itraconazole on the pharmacokinetics of RO7017773 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria

* Healthy (absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology and urinalysis) as judged by the Investigator.
* Male and women of non-childbearing potential (WONCBP)

Exclusion Criteria

* History of convulsions (other than benign febrile convulsions of childhood) including epilepsy, or personal history of significant cerebral trauma or central nervous system (CNS) infections (e.g., meningitis)
* History of clinically significant hypersensitivity or allergic reactions
* Abnormal blood pressure
* Abnormal pulse rate
* History or presence of clinically significant ECG abnormalities before study drug administration or cardiovascular disease
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* Positive test for drugs of abuse or alcohol
* Evidence of human immunodeficiency virus (HIV) infection
* Presence of hepatitis B surface antigen (HBsAg) or positive HCV antibody test result at screening or within 3 months prior to starting study treatment
* Participants who regularly smoke more than 5 cigarettes daily or the equivalent and are unable or unwilling not to smoke during the in-house period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- BIOTRIAL, Rennes, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy male and female participants between 18 and 55 years old. Female participants were women of non-childbearing potential (WONCBP).
Groups:
- RO7017773 Alone, Then RO7017773 + Itraconazole: In Period 1, participants received a single dose of RO7017773 alone in a fed state. In Period 2, participants received a single dose of RO7017773 after repeated doses of itraconazole in a fed state.
Period: Period 1
Arm/Group | RO7017773 Alone, Then RO7017773 + Itraconazole
Started | 14
Completed | 14
Not Completed | 0
Period: Period 2
Arm/Group | RO7017773 Alone, Then RO7017773 + Itraconazole
Started | 14
Completed | 13
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | RO7017773 Alone, Then RO7017773 + Itraconazole
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of RO7017773 in Plasma
Time Frame: Period 1 (RO7017773) and Period 2 (RO7017773 + Itraconazole)
Population: The pharmacokinetic set (PKS) included all participants who received at least one dose of study treatment and who had data from at least one post-dose sample. This outcome measure is specific to the reported arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- RO7017773 Alone: In Period 1, participants received a single dose of RO7017773 alone in a fed state.
- RO7017773 + Itraconazole: In Period 2, participants received a single dose of RO7017773 after repeated doses of itraconazole in a fed state.
Arm/Group | RO7017773 Alone | RO7017773 + Itraconazole
Number analyzed (Participants) | 13 | 13
ng/mL | 458 (32.1) | 516 (22.7)

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: 12 weeks
Population: The safety set (SS) included all participants who received at least one dose of study treatment and included any participant(s) that were withdrawn from the study.
Measure: Number; unit: Percentage of Participants
Groups:
- Itraconazole Alone; RO7017773 + Itraconazole: In Period 2, participants received a single dose of RO7017773 after repeated doses of itraconazole in a fed state.
Arm/Group | RO7017773 Alone | Itraconazole Alone | RO7017773 + Itraconazole
Number analyzed (Participants) | 14 | 14 | 13
Percentage of Participants | 57.1 | 14.3 | 53.8

3. Secondary Outcome: Change in Suicide Risk as Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is an assessment tool to evaluate suicidal ideation and behavior. Categories have binary responses (yes/no) and include: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation or behavior is indicated by a "yes" answer to any of the listed categories. A score of 0 is assigned if no suicide risk is present.
Time Frame: From screening visit through Period 2 Day 11
Population: The included set (IS) contained all study participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | RO7017773 Alone | RO7017773 + Itraconazole
Number analyzed (Participants) | 14 | 13
Units on a scale
  Screening | 0 (0) | 0 (0)
  Period 2 Day 11 | 0 (0) | 0 (0)

4. Secondary Outcome: Cmax of Itraconazole in Plasma
Time Frame: Period 2
Population: The pharmacokinetic set (PKS) included all participants who received at least one dose of study treatment and who had data from at least one post-dose sample. This outcome measure is specific to the reported arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | RO7017773 Alone
Number analyzed (Participants) | 13
ng/mL | 724 (43.2)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | RO7017773 Alone | Itraconazole Alone | RO7017773 + Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 8/14 | 2/14 | 7/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RO7017773 Alone (N=14) | Itraconazole Alone (N=14) | RO7017773 + Itraconazole (N=13)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT03774576/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT03774576/SAP_001.pdf